CLINICAL TRIAL: NCT07043985
Title: Effect of Intraepidermic Injection of Vitamin C on Collagen Production Compared to Fibrotic Hereditary Gingival Fibromatosis: Histopathological Study
Brief Title: Effect of Vitamin C on Collagen Production in Comparison to Hereditary Gingival Fibromatosis: Histopathological Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Badr University (Other)
Collaborators: Cairo University (Other)
Responsible Party: Principal Investigator, Rasha Wagih, assistant professor, Badr University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: BUC-IACUC-250423-130
Record Dates: First submitted 2025-06-17; First posted 2025-06-29 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Tissue Modification After Vit c Injection
MeSH Terms: interventions — Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- G1 (positive control): 5 patients suffering from non-syndromic HGF (Experimental): Gingival bioposy was evaluated
  Interventions: Diagnostic Test: biopsy
- G2 (negative control): 5 patients of normal healthy gingival tissue (negative control) (Experimental): normal healthy gingival tissue biopsy
  Interventions: Diagnostic Test: biopsy
- received intraepidermic vitamin C injection for non-inflammatory purpose (Active Comparator): vit C injection for non-inflammatory purpose
  Interventions: Diagnostic Test: biopsy
- G4: 5 patients received vitamin C injection for inflammatory purposes (Active Comparator): vitamin C injection for inflammatory purposes
  Interventions: Diagnostic Test: biopsy

INTERVENTIONS:
Diagnostic Test: biopsy — Diagnosis of the HGF and healthy tissues depends on pre-described criteria; gingival overgrowth covering one third of the crown length as a minimum, systemically free, no history of drug uptake causing gingival overgrowth (nifedipine, phenytoin, cyclosporine, oral contraceptive pills). Before sampling, written consents were obtained from all patients. Using light microscope, haematoxylin and eosin (H&E) stained sections were precisely examined and histopathological features were reported. All specimens were assessed semi-quantitatively, on a graded scale, under ×100 magnification power and a fixed grid for the following parameters. Three to four fields of each gingival specimen were randomly selected. A blinded evaluation was done by two independent observers. If a debate was reported regarding a specimen, a consensus was reached following re-evaluation. The most representative areas were selected to be morphometrically analyzed using Leica QWin 500 analyzer computer system (Germany).

SUMMARY:
In this preliminary study, we propose that the intraepidermic injection of vit C can induce quantitative and qualitative modification of the gingival biotype. We also propose that such improvement is lacking of any pathologic transformation when will compare to the hereditary gingival fibromatosis with highlighting the mechanism of fibrous tissue formation. The study aims secondly to provide a detailed explanation for the pathogenesis of HGF.

DETAILED DESCRIPTION:
Oral fibromatosis is a benign non-relevant condition that could be an idiopathic solitary manifestation, part of a syndrome or a manifestation associated with systemic disease as leukemia, epilepsy, etc. (Anegundi et al., 2006 and Hakkinen & Csiszar, 2007). It may be also associated with other minor manifestations as hypertrichosis (Pavone, 2015 and Sabina-Pena-Borges, 2015), anemia, gastro-intestinal disturbance and/ or hormonal disturbance. Up till now, the idiopathic form is a rare condition with no definite hypothesis that could explain its mechanism.

Clinically, the disease usually develop as fibrotic non-painful, pinkish, non-hemorrhagic lesions which can either relate to erupted teeth (deciduous or permanent) or edentulous areas (retromolar region, maxillary tuberosity). The lesions primarily erupt as nodular separate islands related to the interproximal papillae then gradually coalesce (Anegundi et al., 2006; Singhal, 2013 and Gawron et al., 2016).

By the development of such lesions, bad esthetics, speech problems, mastication problems, carious lesions, plaque accumulation are the main complaints of the patients suffer from. Bone loss as well as periodontitis may develop later on as a squeal of plaque accumulation and improper cleaning (Ramer et al., 1996 and Anegundi et al., 2006). The peak of enlargement usually accompanies the beginning of mixed dentition (Anegundi et al., 2006; Singhal, 2013 and Gawron et al., 2016).

According to literature, the genetic susceptibility showed the most reliable explanation to fibromatosis development. It may be transmitted as an autosomal dominant or recessive trait. Local factors also play an important role in disease exacerbation such as plaque, calculus, chemical agents, trauma, restorations, orthodontic appliances, fixed restorations (Anegundi et al., 2006).

Histologically, there is great debate if the enlargement's origin is more relevant to epidermis layer, dermis layer or both. In the epidermal theory, the epithelial layer is the initiating layer due to the epithelial mesenchyme transitions and the presence of keratinocyte growth factor (Boukamp et al., 1990) while in the dermal theory, the overproduction of the dense, fibrous and avascular extracellular matrix with differently oriented collagen bundles, marked reduction in collagenase formation are the initiating factors (Vardar et al., 2005; El-Firt, 2011; Pego et al., 2015). The name fibromatosis is related to the dermal hypothesis due to the over production of fibrous tissues. Finally, the coexistence of epithelial and connective tissue hyperplasia regards to fibroblasts and keratinocytes hyperactivity which supports the third theory (Boukamp et al., 1990).

Away from the pathological conditions, gingival thickness could be intentionally induced to modify the oral tissue biotype using vitamin C (vit C), which has antioxidant and anti-inflammatory properties (Yussif et al., 2016). On microscopic examination, vitamin C tissue modification histologically resembles gingival fibromatosis. Therefore, it is quite important to cautiously examine the biotype modification occurs during vitamin C injection.

Gingival tissue biotype exhibits great clinical significance in preserving the gingival health, determining the treatment outcome and the prognosis of periodontal apparatus (Abraham et al., 2014).

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed as HGF
* patients diagnosed with altered passive eruption who needs excess gingival tissue removal
* no age or gender predilection

Exclusion Criteria:

* patienst undertaken drugs cause gingival enlargment
* prednent and lactating mothers

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-01-03 (Actual); Primary Completion 2024-11-05 (Actual); Study Completion 2025-05-06 (Actual)

PRIMARY OUTCOMES:
Area percent occupied by connective tissue | 7
  the percent of the tissues occupied by connective tissue only

SECONDARY OUTCOMES:
Density of Collagen bundles | 7
  the percent amount of the collagen bundles

CONTACTS AND LOCATIONS:
Locations (1):
- Entertainment Area, Badr City, Cairo, Egypt, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided